CLINICAL TRIAL: NCT05929170
Title: Comparison of Different Tipe Extremely Obese Patients Undergoing Gastric Sleeve Surgery in Terms of Perioperative Risk (Cardiopulmonary Parameters and Other Perioperative Risk Factors) and Effectiveness of the Intervention
Brief Title: Comparison of Extremely Obese Patients Undergoing Gastric Sleeve Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Siptár Miklós, Anesthesiologist and ICU specialist, University of Pecs
Other Study IDs: 8653-PTE 2021.
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Morbid; Hypertension; Diabetes Mellitus, Type 2
Keywords: gastric sleeve operation
MeSH Terms: conditions — Obesity, Morbid; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By the comparison of the preoperative and postoperative data of approximately 160 patients undergoing gastric sleeve surgery, we try to draw conclusions about the effectiveness of gastric sleeve surgery, expected complication rate.

DETAILED DESCRIPTION:
We plan to compare the preoperative and postoperative data of approximately 160 patients undergoing gastric sleeve surgery (android-gynoid, male-female, comparison of patients with different degree of obesity, age comparison, etc.) Many preoperative and postoperative data are known about the patients (weight, height, BMI, preoperative comorbidities, heart ultrasound values, respiratory function values, laboratory parameters, smoking habits, rate of weight loss in half a year and one year, etc.). By statistical analysis of these data, we try to draw conclusions about the effectiveness of gastric sleeve surgery, expected complication rate, etc.,

ELIGIBILITY:
Inclusion Criteria:

Obesity (BMI higher than 30 kg/m2)

Exclusion Criteria:

Lack of patient consent to the study, Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients (BMI Higher than 30 kg/m2)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assessing the results of gastric sleeve surgery, by weight loss | up to one year
  weight loss (kg)

SECONDARY OUTCOMES:
Assessing the half and one-year results of gastric sleeve surgery, by change in comorbidities | half year, one year
  change in comorbidities (the clinical improvement of the given comorbidity, for example in the case of hypertension, the patient's antihypertensive medications can be reduced or completely omitted, ect.)
Assessing the half and one-year results of gastric sleeve surgery, comparing different groups (male-female, android-gynoid tipe of obesity, ect.) | half year, one year
  weight loss (kg)
Assessing the half and one-year results of gastric sleeve surgery, weight loss. (We try to find a confluence between the perioperative parameters and the expected outcome) | half year, one year
  weight loss (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Siptár Miklós, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No